CLINICAL TRIAL: NCT01398436
Title: Comparison Between Hemoglobin Saturation in the Superior Vena Cava and in the Right Atrium
Brief Title: Hemoglobin Saturation in Superior Vena Cava and Right Atrium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Franco Cavaliere, Associate Professor of Anaesthesia and Intensive Care, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: P/999/CE/2010
Record Dates: First submitted 2011-07-19; First posted 2011-07-20 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2013-04

CONDITIONS: Cardiac Surgery; Shock
Keywords: Central venous saturation; Mixed venous saturation; Right atrium; Central Venous Catheter position
MeSH Terms: conditions — Shock

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Catheter tip in right atrium (Experimental): In this group a central venous catheter will be advanced for its entire length unless arrhythmias develop.Catheter position will be controlled by transesophageal echocardiography and/or by chest radiography.
  Interventions: Procedure: central venous catheter positioning in right atrium
- Catheter tip in superior vena cava (No Intervention): In this group a central venous catheter will be inserted for 15 cm in accordance with standard practice. Catheter position will be controlled by transesophageal echocardiography and/or by chest radiography

INTERVENTIONS:
Procedure: central venous catheter positioning in right atrium — A central venous catheter will be advanced for its entire length unless arrhythmias develop. Catheter position will be controlled by transesophageal echocardiography and/or by chest radiography
  Arms: Catheter tip in right atrium

SUMMARY:
The aim of the study is to compare oxygen saturation of blood samples collected from the superior vena cava, the right atrium, and the pulmonary artery. A secondary target was to assess whether positioning the tip of central venous catheters in the right atrium causes more arrhythmias than positioning it in the superior vena cava.

The study is carried out in patients that undergo central venous and pulmonary artery catheterization for surgical coronary revascularization. In the interventional group (atrium, A), the tip of the central venous catheter (CVC) is placed in the right atrium; in the control group (control, C), the tip is placed in the superior vena cava. In both groups, CVC position is confirmed with transesophageal echocardiography (TEE). At fixed times during surgery and in the following 72 hours, heparinized blood samples are collected from the proximal and distal CVC lumens and from the distal lumen of the pulmonary catheter (PC) and oxygen saturation is measured by an oximeter. Besides, mechanical and electrical complications potentially influenced by CVC position are registered.

1. The primary aim of the study will be achieved by performing the following analysis on values from CVC proximal and distal lumens:

   1. a Bland Altman analysis between proximal and distal oxygen saturation in group A, in order to evaluate if the two measures are equivalent
   2. a comparison of the difference between proximal and distal oxygen saturation in groups A and C in order to rule out random errors
2. In addition:

   1. differences in oxygen saturation between proximal or distal CVC and distal PC will be compared in order to evaluate whether distal saturation is more indicative of mixed venous saturation
   2. differences between proximal and distal oxygen saturation will be correlated with cardiac index and PCWP to investigate if low cardiac output and hypovolemia increase differences
3. The secondary aim of the study will be achieved by comparing the incidence of cardiac arrhythmias in groups A and C

DETAILED DESCRIPTION:
The study design is a prospective, randomized, open-label study. Forty consecutive patients undergoing cardiac surgery requiring the placement of a central venous catheter and of a Swan-Ganz catheter, and then admitted to Cardiac Surgery ICU of "A.Gemelli" University Hospital will be included in the study. Patients will be randomized to two groups: A group, in which the catheter tip will be positioned in right atrium, and C (control) group, in which the catheter tip will be positioned in the superior vena cava, at the junction with the atrium.

Arrow catheters (3 lumen, 8,5 Fr, 20 cm long) will be used. Catheters will be placed in right internal jugular or subclavian vein with Seldinger technique. In group A, the catheter will be advanced for its entire length unless arrhythmias develop; in group C the catheter will be inserted for 15 cm. Catheter position will be controlled by transesophageal echocardiography and/or by chest radiography. In order to avoid risk of damage to the atrial wall, ECG and central venous pressure will be monitored during the entire observation period, and the catheter will be repositioned, withdrawing it, in presence of extrasystoles or other arrhythmias potentially triggered by contact between the catheter tip and the heart wall, in case of flattening of the curve of the central venous pressure (caused by contact with the atrial wall) or in presence of a ventricular type of curve (migration of the catheter in the right ventricle through the tricuspid valve). The catheter tip will be removed or repositioned in superior vena cava at the time of mobilization of the patient or of his transfer to another unit.

A sample of arterial blood from an arterial line, one of mixed venous blood from the pulmonary catheter and two samples from the CVC, one from the distal lumen and a proximal lumen, will be taken at different times: time 1, at CVC placement; time 2, after sternotomy; time 3, after after discontinuation of CBP; time 4, at admission to ICU; time 5, 6,7 8, respectively 6, 18, 30 and 42 hours after the end of surgery. Samples volume of 1 mL will be collected in heparinized syringes and immediately analyzed by a stat analyzer (Stat Profile Critical Care Xpress by Nova Biomedical) with integrated on-board CO-Oximetry, allowing direct measurement of oxygen saturation.

The values of pH, pO2, pCO2 and saturation of venous samples will be compared and the difference will be analyzed by Bland-Altman method. The observed difference will also be correlated with indexes of tissue perfusion (arterial base excess, arterial plasma lactate) and with the presence and dose of vasoactive drugs infusion.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing cardiac surgery requiring the placement of a central venous catheter and of a pulmonary artery catheter, and then admitted to Cardiac Surgery ICU

Exclusion Criteria:

* age less than 18 years,
* contraindication to catheterization through the right internal jugular or right subclavian vein
* presence of inflammatory disease of the heart (eg myocarditis) or any other disease increasing the risk of complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2011-03; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Difference between oxygen saturation in blood collected from the proximal and distal lumens of a central venous catheter the tip of which is positioned in the right atrium | 72 hours
  Large differences from the proximal and distal lumens means that blood from the superior vena cava is poorly representative of blood from the inferior vena cava and the coronary sinus
Difference between oxygen saturation | 72 hours
  Difference between oxygen saturation in blood collected from the proximal and distal lumens of a central venous catheter the tip of which is positioned in the right atrium and oxygen saturation in pulmonary artery

SECONDARY OUTCOMES:
Safety of central venous catheters with the tip in the right atrium in ICU patients | 72 hours
  To evaluate the incidence of arrhythmic and traumatic complications in the study group and in controls

CONTACTS AND LOCATIONS:
Overall Officials: Franco Cavaliere, Professor, Principal Investigator — Catholic University of Sacred Heart, Rome
Locations (1):
- Università Cattolica del Sacro Cuore - Policlinico "A. Gemelli", Rome, Italy

REFERENCES:
- [Background] Dueck MH, Klimek M, Appenrodt S, Weigand C, Boerner U. Trends but not individual values of central venous oxygen saturation agree with mixed venous oxygen saturation during varying hemodynamic conditions. Anesthesiology. 2005 Aug;103(2):249-57. doi: 10.1097/00000542-200508000-00007. PMID 16052106
- [Background] Edwards JD, Mayall RM. Importance of the sampling site for measurement of mixed venous oxygen saturation in shock. Crit Care Med. 1998 Aug;26(8):1356-60. doi: 10.1097/00003246-199808000-00020. PMID 9710094
- [Background] Chawla LS, Zia H, Gutierrez G, Katz NM, Seneff MG, Shah M. Lack of equivalence between central and mixed venous oxygen saturation. Chest. 2004 Dec;126(6):1891-6. doi: 10.1378/chest.126.6.1891. PMID 15596689
- [Background] Pikwer A, Baath L, Davidson B, Perstoft I, Akeson J. The incidence and risk of central venous catheter malpositioning: a prospective cohort study in 1619 patients. Anaesth Intensive Care. 2008 Jan;36(1):30-7. doi: 10.1177/0310057X0803600106. PMID 18326129
- [Background] Webster CS, Merry AF, Emmens DJ, Van Cotthem IC, Holland RL. A prospective clinical audit of central venous catheter use and complications in 1000 consecutive patients. Anaesth Intensive Care. 2003 Feb;31(1):80-6. doi: 10.1177/0310057X0303100116. PMID 12635401
- [Derived] Cavaliere F, Zamparelli R, Martinelli L, Scapigliati A, De Paulis S, Caricato A, Gargaruti R, Cina A. Blood from the right atrium may provide closer estimates of mixed venous saturation than blood from the superior vena cava. A pilot study. Minerva Anestesiol. 2014 Jan;80(1):11-8. Epub 2013 Jul 15. PMID 23857438